CLINICAL TRIAL: NCT02478437
Title: A Prospective Trial of Cooled Radiofrequency Ablation of Medial Branch Nerves for the Treatment of Lumbar Facet Syndrome
Brief Title: A Trial of Cooled Radiofrequency Ablation of Medial Branch Nerves for theTreatment of Lumbar Facet Syndrome
Acronym: STU00097239
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Pain Society (Other)
Responsible Party: Principal Investigator, David Walega, Associate Professor, Chief, Division of Pain Medicine, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU00097239
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
Keywords: Lumbar Facet Syndrome
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Conventional radiofrequency ablation (RFA) Following ablation, 0.5 cc of 0.5% bupivacaine will be injected to provide post procedure analgesia.
  Interventions: Procedure: Conventional radiofrequency ablation (RFA)
- Group 2 (Active Comparator): Cooled radiofrequency ablation (CRFA) Following ablation, 0.5 cc of 0.5% bupivacaine will be injected to provide post procedure analgesia.
  Interventions: Procedure: Cooled Radiofrequency Ablation (CRFA)

INTERVENTIONS:
Procedure: Conventional radiofrequency ablation (RFA) — A conventional RFA electrode with a 10mm active tip will be used. RFA lesions will be performed for 90 seconds with the maximum electrode temperature raised to 80°C.
  Arms: Group 1
Procedure: Cooled Radiofrequency Ablation (CRFA) — Following 18G C-RFA electrode positioning, 1cc of 2% lidocaine will be injected through the introducer needle for anesthesia during the ablation. The maximum electrode temperature is 60°C.
  Arms: Group 2

SUMMARY:
This study is being done to determine whether cooled radiofrequency ablation (CRFA) on the medial branch nerves of the lumbar facet joint is effective for the treatment of low back pain. CRFA blocks the nerves that carry pain signals from joints in the lower back such that the brain does not receive the message that the low back is in pain. This technique is commonly performed by burning these nerves rather freezing them, but it is suspected that freezing them results in better pain relief. The CRFA blocks has been shown to effectively treat sacroiliac joint pain (a joint in the pelvis), which is another reason that it is suspected that CRFA will be effective when treating pain related to facet joints in the low back. We are performing this study in order to determine if that is the case.

DETAILED DESCRIPTION:
The CRFA blocks has been shown to effectively treat sacroiliac joint pain (a joint in the pelvis), which is another reason that it is suspected that CRFA will be effective when treating pain related to facet joints in the low back. We are performing this study in order to determine if that is the case.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar facet syndrome pain who would undergo treatment by lumbar medial branch radiofrequency ablation.
* Low back pain for at least 6 months.
* Pain resistant to conventional therapy including NSAIDs, opioids, muscle relaxants, oral steroids, physical therapy or chiropractic care.
* Pain diagram suggesting possibility of facet-mediated pain.
* Referred pain when present not beyond the knee.
* Positive response to at least 1 set of diagnostic intra-articular facet injections or medial branch blocks, defined as > 75% reduction in pain following diagnostic blocks with local anesthetic (0.5mL of 0.5% bupivacaine OR 0.5 mL of 2% lidocaine).

Exclusion Criteria:

* Focal neurologic signs or symptoms.
* Radiologic evidence of a symptomatic herniated disc or nerve root impingement related to spinal stenosis.
* Previous radiofrequency ablation treatment for similar symptoms.
* Patient refusal.
* Lack of consent.
* Active systemic or local infections at the site of proposed needle and electrode placement.
* Coagulopathy or other bleeding disorder, current use of anticoagulants or anti-platelet medications.
* Allergy to medications being used for injection procedures (contrast dye, local anesthetic, IV sedative).
* Inability to read English, communicate with staff, or participate in follow up.
* Pregnancy.
* Cognitive deficit.
* Negative response to diagnostic intra-articular facet injections or medial branch blocks, defined as < 75% reduction in pain following diagnostic blocks with local anesthetic (0.5mL of 0.5% bupivacaine OR 0.5 mL of 2% lidocaine).
* Daily opiate analgesic use more exceeding 3 months prior to study inclusion.
* Unstable medical or psychiatric illness.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Pain improvement | 6 months post-procedure
  Percent of participants who reported 50% or greater improvement in pain

SECONDARY OUTCOMES:
Global pain score | 1 month, 3 months, 6 months and 12 months post procedure
  Global Numeric Rating Scale (NRS, 0 is no pain and 10 is worst pain imaginable)
McGill Pain Questionnaire (MPQ) | 1 month, 3 months, 6 months and 12 months post procedure
  Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain).
Pain Anxiety Symptom Scale short form (PASS-20) | 1 month, 3 months, 6 months and 12 months post procedure
  The PASS-20 assesses 4 factorially distinct components of pain-related anxiety. Each question is in a form of a 6-point Likert Scale anchored from 0 (never) to 5 (always).
Center for Epidemiologic Studies Depression short form index (CESD-10) | 1 month, 3 months, 6 months and 12 months post procedure
  The possible range of the 10-item scale is 0 to 30, and a cut off score of ten or higher indicates the presence of significant depressive symptoms. Subjects responded to each item of the scale by rating the frequency of each mood or symptom ''during the past week'' on a four-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Anesthesiology Pain Managment Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCormick ZL, Choi H, Reddy R, Syed RH, Bhave M, Kendall MC, Khan D, Nagpal G, Teramoto M, Walega DR. Randomized prospective trial of cooled versus traditional radiofrequency ablation of the medial branch nerves for the treatment of lumbar facet joint pain. Reg Anesth Pain Med. 2019 Mar;44(3):389-397. doi: 10.1136/rapm-2018-000035. PMID 30777903